CLINICAL TRIAL: NCT05322304
Title: Randomized Controlled Trial of Almond Supplementation vs. Isocaloric Diet on Cognitive Functions in Middle-aged (40-60 Years) Asian Indians With Prediabetes
Brief Title: Almonds and Cognitive Functions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diabetes Foundation, India (Other)
Collaborators: National Diabetes Obesity and Cholesterol Foundation (Other); Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NDOC.12/2022
Record Dates: First submitted 2022-03-25; First posted 2022-04-11 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: PreDiabetes
Keywords: almonds; prediabetes; cognition
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: parallel arm randomized controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- almond (Experimental): dietary intervention with almonds ()20% of energy)
  Interventions: Dietary Supplement: Almond
- Control (No Intervention): usual diet and lifestyle

INTERVENTIONS:
Dietary Supplement: Almond — Intervention (almond supplementation) and Isocaloric diets (control)
  Arms: almond

SUMMARY:
Initial Recruitment and Sensitization: In this free-living randomized control parallel arm study of 24 weeks of almond intervention, we shall recruit apparently healthy middle aged (age range 40-60 years)prediabetic Asian Indians having fasting blood glucose ≥100mg/dl and <126 mg/dl and /or 2-h plasma glucose ≥140mg/dl and <200mg/dl (after ingestion of 75-gram anhydrous oral glucose).

DETAILED DESCRIPTION:
Objectives and Measurements:

a. Primary Objective: To evaluate the effect of almond supplementation on cognitive functions Co-primary Objective: To evaluate changes in neuroimaging (blood flow, and the expression of functional brain networks during cognitive demands) using functional MRI.

Flow of Study Procedures

1. This will be a randomized controlled parallel arm study on free living Asian Indians, selected based on inclusion criteria.
2. Sample size: 60 (n, 30 in each arm)
3. After recruitment subjects would enter the run-in period for 2 weeks when they would be given standard diet and lifestyle modification counseling formulated according to guidelines for Asian Indians.
4. Subjects would be screened again just for inclusion/exclusion criteria at the end of the run-in period and would be randomized either to the experimental group or control group
5. Composition of diets:

   i. Intervention group: Individualized diets incorporating almonds, 20% energy. Macronutrient composition: Carbohydrates,49%en., fats,32%en., and proteins, 19%en.

   ii. Control group: Isocaloric diet. Macronutrient composition: Carbohydrates,50%en., fats, 35%en., proteins,15%en.
6. The diet (as above) and lifestyle modification will be continued in both groups for 6 months with rigorous compliance
7. Compliance Checks: The diet (as above) and lifestyle modification will be continued in both groups for 6 months with rigorous compliance check .

Compliance for the intervention in all the subjects (control and intervention group) will be checked by taking following measures:

1. Biweekly telephonic calls. During these telephonic calls compliance to diet, exercise, almond intake, adverse event or any problem with the intervention will be assessed. Calls will be recorded in a call log and subject compliance (consumption of almonds) will be recorded in the proforma.
2. Text messages reminding intake of almonds (weekly) and face-to-face interactions (once every month, at least 20 min each session) discussing problems if any.

ELIGIBILITY:
Inclusion Criteria:

1. Asian Indians having fasting blood glucose ≥100mg/dl and <126 mg/dl and /or 2-h plasma glucose ≥140mg/dl and <200mg/dl (after ingestion of 75-gram anhydrous oral glucose)
2. age 40-60 years

Exclusion Criteria:

1. Subjects Having Inability to Undergo Neuropsychological Testing
2. Previously Diagnosed Neurodegenerative Disease Prior Stroke
3. Significant Head Trauma, or Brain Surgery
4. Relevant Psychiatric Illness
5. Major Depression
6. Morbid Obesity
7. Diabetes
8. Uncontrolled Hypertension
9. Prior Chemotherapy
10. Allergy to Almonds
11. Habitual Consumption of Tree nuts (>2 Servings/Wk.); or Customary Use Of Fish Oil, Flaxseed Oil, and/ Or Soy Lecithin
12. Chronic Smoking
13. Alcohol abuse (> 2 Drinks, 60 Ml Of Whisky Per Day)
14. Severe Dyslipidemia (Total Cholesterol > 300 Mg/Dl, Serum Triglycerides > 500mg/Dl)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
neuropsychological function | 2 year
  cognitive functions using computerized neuropsychological assessment systems (CANTAB

CONTACTS AND LOCATIONS:
Locations (1):
- National Diabetes Obesity and cholesterol Foundation (NDOC), Delhi, India